CLINICAL TRIAL: NCT00191048
Title: Open-Label Treatment With Atomoxetine Hydrochloride in Child and Adolescents With Attention-Deficit/Hyperactivity Disorder and Comorbid Dyslexia
Brief Title: Treatment With Atomoxetine Hydrochloride in Children and Adolescents With ADHD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7975; B4Z-US-LYCE
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-01-26 (Estimated); Status verified 2007-01

CONDITIONS: Attention-Deficit/Hyperactivity Disorder; Comorbid Dyslexia
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride

INTERVENTIONS:
Drug: Atomoxetine

SUMMARY:
The purpose of this study is to assess the efficacy and safety of atomoxetine administered once daily in the treatment of children and adolescents with ADHD and comorbid dyslexia.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ADHD only or ADHD and Dyslexia
* At least 10 years old and no more than 16 years old
* IQ score of 80 or more
* Must be able to swallow capsules

Exclusion Criteria:

* Have received treatment within last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry
* Weigh less than 25 kg or greater than 70 kg
* Pregnant or breast feeding
* Documented history of bipolar I or II disorder, or psychosis
* Documented history of autism, Asperger's syndrome or pervasive developmental disorder

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 105
Dates: Start 2003-10; Study Completion 2006-03

PRIMARY OUTCOMES:
To assess the effect of atomoxetine,given for approximately 16 weeks, in the treatment of ADHD with Dyslexia as measured by the ADHDRS-IV-Parent:Inv

SECONDARY OUTCOMES:
To assess the effect of atomoxetine on educational testing, working memory,and adaptive functioning throughout 16 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (8):
- United States (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Rolling Hills Estate, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Maitland, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Libertyville, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Las Vegas, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Oklahoma City, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Nashville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Burlington, Vermont

REFERENCES:
- [Derived] Sumner CR, Gathercole S, Greenbaum M, Rubin R, Williams D, Hollandbeck M, Wietecha L. Atomoxetine for the treatment of attention-deficit/hyperactivity disorder (ADHD) in children with ADHD and dyslexia. Child Adolesc Psychiatry Ment Health. 2009 Dec 15;3:40. doi: 10.1186/1753-2000-3-40. PMID 20003507